CLINICAL TRIAL: NCT00158964
Title: EASYTRAK® 4 STEERABLE LV Lead Clinical Investigation
Brief Title: EASYTRAK 4 Steerable LV Lead
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Clinicals0006
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-06-25 (Estimated); Status verified 2007-06

CONDITIONS: Heart Failure
Keywords: left ventricular lead; pacing; heart failure
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Device: EASYTRAK 4 STEERABLE LV lead

SUMMARY:
The primary objective of this clinical investigation is to evaluate the safety and effectiveness of the EASYTRAK 4 STEERABLE LV lead.

DETAILED DESCRIPTION:
This is a prospective, multi-center clinical study is to evaluate the safety and effectiveness of the EASYTRAK 4 STEERABLE LV lead.

ELIGIBILITY:
Inclusion Criteria:

* Must receive a commercially available Guidant CRT-P or CRT-D device
* Creatinine < 2.5 mg/dL obtained no more than two weeks prior to enrollment
* Age 18 or above, or of legal age to give informed consent specific to state and national law
* Willing and capable of providing informed consent, undergoing a device implant, participating in all testing associated with this clinical investigation at an approved clinical investigation center and at the intervals defined by this protocol
* Geographically stable residents who are available for follow-up

Exclusion Criteria:

* Have a known hypersensitivity to a 1.0 mg (0.5 mg per electrode) nominal dose of dexamethasone acetate
* Have or had previous cardiac resynchronization therapy, a coronary venous pace/sense lead or attempted LV lead placement
* Have pre-existing cardioversion/defibrillation leads or right ventricular pacing leads other than those specified in the investigational plan (unless the investigator intends to replace them with permitted cardioversion/defibrillation leads)
* Currently requiring dialysis
* Have had a myocardial infarct, unstable angina, percutaneous coronary intervention, or coronary artery bypass graft during the preceding 30 days prior to enrollment
* Have hypertrophic obstructive cardiomyopathy or infiltrative cardiomyopathy (e.g., amyloidosis, sarcoidosis)
* Documented life expectancy of less than six months or expected to undergo heart transplant within the next six months
* Enrolled or participating in any concurrent study, including drug investigations, without Guidant written approval, that may confound the results of this study
* Have a pre-existing unipolar pacemaker that will not be explanted/abandoned
* Have a mechanical tricuspid heart valve
* Women who are pregnant or plan to become pregnant Note: Women of childbearing potential must have a negative pregnancy test within seven days of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2005-03; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Lead-related complication free-rate at 3-months.
Chronic mean pacing thresholds at 3-months.

SECONDARY OUTCOMES:
Chronic Mean pacing impedances at 3-months
Chronic Mean R-wave amplitudes at 3-months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Mester, MD, Principal Investigator — Tampa General Hospital
Locations (1):
- Multiple locations, Saint Paul, Minnesota, United States